CLINICAL TRIAL: NCT00993577
Title: Global Postural Reeducation and Static Stretching Exercises in the Treatment of Myogenic Temporomandibular Disorders. A Randomized Study
Brief Title: Stretching Exercises and Temporomandibular Disorders
Acronym: Stretching
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Amelia Pasqual Marques, FMUSP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 155/04
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Temporomandibular Disorders
Keywords: Stretching; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Muscle Stretching Exercises; Exercise Therapy; Pain Measurement; Arthrocentesis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercises (Experimental): Global Postural Reeducation Static Stretching Exercises
  Interventions: Other: Stretching exercises; Device: Stretching exercises; Device: Exercises

INTERVENTIONS:
Other: Stretching exercises — Treatment consisted of eight individual sessions (once a week), over two months. At the first 10 minutes of sessions, patients rested (supine position) with all limbs relaxed. Manual therapy maneuvers were made as described by Bienfait,17 associated to breathing exercises, in order to stretch the fasciae that recover the shoulders, as well as the cervical spine muscles. After that, stretching treatment (global or static) was conducted for another 30 minutes.
  Other Names: Global Postural Reeducation; Static Stretching Exercises
Device: Stretching exercises — Treatment consisted of eight individual sessions (once a week), over two months. At the first 10 minutes of sessions, patients rested (supine position) with all limbs relaxed. Manual therapy maneuvers were made as described by Bienfait,17 associated to breathing exercises, in order to stretch the fasciae that recover the shoulders, as well as the cervical spine muscles. After that, stretching treatment (global or static) was conducted for another 30 minutes.
  Other Names: Global Postural Reeducation; Static Stretching Exercises
Device: Exercises — Treatment consisted of eight individual sessions (once a week), over two months. At the first 10 minutes of sessions, patients rested (supine position) with all limbs relaxed. Manual therapy maneuvers were made as described by Bienfait,17 associated to breathing exercises, in order to stretch the fasciae that recover the shoulders, as well as the cervical spine muscles. After that, stretching treatment (global or static) was conducted for another 30 minutes.
  Other Names: Muscle stretching exercises; Pain measurement; Temporomandibular joint.

SUMMARY:
To compare the efficacy of global postural reeducation (GPR) with static stretching exercises (SS) in the treatment of women with temporomandibular disorders (TMD).

Physical therapy is of importance in the treatment of myogenic temporomandibular disorders (TMD). Both stretching exercise and global posture reeducation are equally effective in the treatment of TMD.

DETAILED DESCRIPTION:
Purpose: To compare the efficacy of global postural reeducation (GPR) with static stretching exercises (SS) in the treatment of women with temporomandibular disorders (TMD).

Methods: A total of 24 subjects with TMD were randomized into two treatment groups: GPR, where therapy involved muscle global chain stretching, or SS, with conventional static stretching. Eight treatment sessions lasting 40 minutes each (weekly) were performed. Assessments were conducted at baseline, immediately after treatment end, and again two months later. Measurements included pain intensity at the temporomandibular joint, headache, cervicalgia (visual analogue scale - VAS) and teeth clenching. Additionally, electromyographic activity and pain thresholds were measured at the masseter, anterior temporalis, sternocleidomastoid, and upper trapezius muscles. Two-way analysis of variance (ANOVA) with Tukey post-hoc test was used for in-between group comparisons. Significance level was 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Helkimo index III,
* Myogenic TMD, AND
* Presence of para-functional habits, such as: bruxism, teeth clenching, mouth-breathing and lip biting.

Exclusion Criteria:

* Surgery or trauma in the orofacial region,
* Systemic or degenerative diseases, OR
* Undergoing odontological, psychological, or physical therapy treatments.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-02; Primary Completion 2006-07 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Pain | 2

SECONDARY OUTCOMES:
Quality of life | 2

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Physicaltherapy, Speech and Ocupational Therapy Department, Rua Cipotânea, 51, São Paulo
  - Clinical Hospital of University of São Paulo, São Paulo, São Paulo